CLINICAL TRIAL: NCT00675974
Title: Prospective Randomized Study of the Effectiveness of Prospective Randomized Study on the Effectiveness of Pressure Garment Therapy for the Prevention of Hypertrophic Scarring in Burned Children
Brief Title: Use of Pressure Garments for Burn Scars
Acronym: Jobst
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-126; NIDRR
Record Dates: First submitted 2007-12-26; First posted 2008-05-12 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Burns
Keywords: Burn; Scar; Pressure garments; Wound healing; Burn Injury
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pressure garment therapy
  Interventions: Device: Jobst Pressure Garment; Device: Medical Z pressure garment
- 2 (No Intervention): No pressure garment therapy

INTERVENTIONS:
Device: Jobst Pressure Garment — Pressure garment therapy for 18 months post burn injury. May be Jobst pressure garment or Medical Z pressure garment.
  Other Names: Jobst pressure garments; Medical Z pressure garments; Pressure garments
  Arms: 1
Device: Medical Z pressure garment — Pressure garment to be worn for 18 months post burn. May be Jobst pressure garment or Medical Z pressure garment.
  Other Names: Pressure garment; Jobst pressure garment
  Arms: 1

SUMMARY:
1. Will Pressure Garment Therapy better control hypertrophic scarring than no Pressure Garment Therapy.
2. How will Pressure Garment Therapy affect functional capacity or scar contracture development across joints either in number or severity.
3. Will Pressure Garment Therapy diminish discomfort due to pruritus.

ELIGIBILITY:
Inclusion Criteria:

* At least 30% total body surface area(TBSA) second degree burns or at least 10% TBSA full-thickness burns including bilateral comparable burns to upper and/or lower extremities.
* at least 1 year of age and no more than 17 years of age
* Wound closure
* No evidence of deep venous thrombosis or other vascular compromise.
* No concomitant conflicting study protocols.

Exclusion Criteria:

* Burn injuries not bilateral to upper and/or lower extremities.
* Evidence of vascular compromise.
* Conflicting protocols.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2012-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Differences in scarring between pressure garment therapy and no pressure garment therapy | Time of burn to 2 years post burn

SECONDARY OUTCOMES:
Effect of Pressure Garment Therapy on functional capacity or scar contracture development across joints either in number or severity compared to no pressure garment therapy. | Time of burn to 2 years post burn
Effect of pressure garment therapy on scar discomfort and pruritis compared to no pressure garment therapy | Time of burn to 2 years post burn

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas